CLINICAL TRIAL: NCT06992258
Title: A Randomized Phase 2 Trial of Fruquintinib and TAS-102 as Compared to Fruquintinib in Patients With Refractory Advanced/Metastatic Colorectal Cancer
Acronym: FRUITION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Criterium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR-AGICC-Fruq-004
Record Dates: First submitted 2025-04-30; First posted 2025-05-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil; HMPL-013

STUDY DESIGN:
Intervention Model Description: Randomized Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fruquintinib and Lonsurf (Experimental)
  Interventions: Drug: Fruquintinib+ Lonsurf (trifluridine and tipiracil)
- Fruquintinib (Active Comparator)
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib+ Lonsurf (trifluridine and tipiracil) — Experimental arm
  Arms: Fruquintinib and Lonsurf
Drug: Fruquintinib — Standard Of Care Arm
  Arms: Fruquintinib

SUMMARY:
A Randomized Phase 2 Trial of Fruquintinib and TAS-102 as Compared to Fruquintinib in Patients with Refractory Advanced/Metastatic Microsatellite Stable Colorectal Cancer

ELIGIBILITY:
1. Provision to sign and date the consent form
2. Able to comply with all study procedures and be available for the duration of the study in the investigator's judgment
3. Age ≥18
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
5. Histologically or cytologically confirmed advanced or metastatic colorectal adenocarcinoma
6. Prior treatment with fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab (unless contraindicated) and cetuximab/panitumumab (for RAS-wild type disease) for the treatment of advanced or metastatic colorectal cancer and had demonstrated progressive disease or intolerance to their last regimen.

   1. Patients who progressed on irinotecan- and oxaliplatin-based regimens previously for metastatic disease should not be retreated with these agents prior to enrolling on this study.
   2. Patients who developed locally advanced/metastatic disease during or within 6 months of completing adjuvant therapy are eligible and the adjuvant/neoadjuvant therapy can be counted as one regimen of chemotherapy for advanced disease. Patients who developed locally advanced/metastatic disease > 6 months after completion of adjuvant therapy must be treated with the above therapies in the advanced setting to be eligible.
7. Mismatch repair proficient (MMRp) status documented by local IHC testing
8. RAS and BRAF status documented
9. Measurable disease according to RECIST v1.1
10. Able to swallow and absorb oral medication
11. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 72 hours prior to first dose of study drug treatment:

    1. ANC ≥ 1.5 × 109/L
    2. Platelet count ≥ 70 × 109/L
    3. Hemoglobin ≥ 9 g/dL in the previous week
    4. Serum bilirubin ≤ 1.5 x the upper limit of normal (ULN); patients with known Gilbert's disease may have a bilirubin ≤ 3.0 ×ULN
    5. Aspartate aminotransferase (AST) and alanine aminotransferase ALT) < 3 × upper limit of normal (ULN) (in the presence of liver metastases ≤ 5 × ULN)
    6. Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault Equation (or similar formula) or as calculated using a timed urine collection
12. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use of contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 180 days after the last study treatment. A woman is considered to be of childbearing potential if she is post-menarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
13. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 180 days after the last dose of study treatment. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion criteria:

1. Patients with known MSI-high or mismatch repair deficient (dMMR) status or in whom the status of both are unknown
2. Patients with BRAF V600 mutations
3. Prior treatment with regorafenib, trifluridine-tipiracil (TAS-102), or fruquintinib.
4. Major surgery within 14 days of C1D1. Minor procedures (e.g. biopsies, central venous catheters) are not considered major surgery.
5. Patients must have recovered from clinically significant AEs of their most recent prior therapy/intervention prior to enrollment as determined by relevant clinical and laboratory parameters.
6. Untreated CNS metastases or known leptomeningeal disease. Patients with treated CNS metastases (either by surgical or radiation techniques) are eligible provided there is no evidence of progression for at least 4 weeks after CNS-directed therapy as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
7. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessments of the investigational regimen. Patients whose prior or concurrent malignancy natural history and/or treatment does NOT have the potential to impact safety or study assessments are eligible.
8. Uncontrolled intercurrent illness (defined as but not limited to others in the opinion of the treating investigator):

   1. Uncontrolled pleural effusion, pericardial effusion or ascites defined as requiring recurrent drainage procedures within 3 weeks of C1D1
   2. Uncontrolled arrhythmia or any ventricular arrhythmia requiring treatment
   3. Uncontrolled hypertension (≥ 160 mmHg systolic or ≥ 100mmHg diastolic in spite of maximal medical therapy)
   4. Urine dipstick or urinalysis with protein ≥ 2+ or 24-hour urine protein ≥ 1.0g/24 hours. Patients with 1+ proteinuria must undergo a urine protein creatinine ratio (UPCR) or 24-hour urine collection to assess protein level. For interpretation of lab values for proteinuria please see Appendix E.
   5. New York Heart Association (NYHA) Functional Classification class 3 or 4 congestive heart failure or left ventricular ejection fraction < 50%
   6. Severe or unstable angina within 3 months prior to C1D1
   7. Active infection requiring IV antibiotics within 1 week prior to C1D1. Antibiotics used for prophylactic purposes are allowed.
   8. Corrected QT interval using the Fridericia method > 470 msec (repeated demonstration of the QTcF interval if > 470 msec during first assessment) or any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as congenital long QT syndrome or family history of long QT syndrome
9. History of or active gastric/duodenal ulcer or ulcerative colitis, active hemorrhage of an unresected gastrointestinal tumor, history of obstruction, perforation or fistulas, and any other condition that could, in the investigator's judgment, result in significant gastrointestinal hemorrhage or perforation, within 6 months prior to C1D1.
10. History or presence of hemorrhage from any other site (e.g. hemoptysis or hematemesis) within 3 months prior to C1D1.
11. History of a venous thromboembolic event (e.g. deep vein thrombosis or pulmonary embolism) within 3 months prior to C1D1.
12. History of an arterial thromboembolic event (e.g. stroke/CVA, transient ischemic event, unstable angina, acute myocardial infarction/coronary artery bypass surgery) within 6 months prior to C1D1.
13. Tumor invasion of a large vascular structure (e.g. pulmonary artery, superior or inferior vena cava).
14. Inability to discontinue medications with a known risk of causing QT prolongation and/or torsades de pointes within 7 days of C1D1.
15. Use of strong or moderate inducers of CYP3A within 7 days of C1D1.
16. Patients with AIDS. HIV-infected patients on effective anti-retroviral therapy with an undetectable viral load during the screening period are eligible.
17. For patients with known chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy during the screening period. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load during the screening period.
18. Recent COVID-19 diagnosis (symptomatic or asymptomatic). To become eligible (following symptomatic infection), the patient must not have fever for 24 hours (without using medicine to reduce fever), other symptoms have improved, and at least 10 days have passed since onset of symptoms. To become eligible (following asymptomatic infection, e.g. positive test only), at least 10 days have passed since the positive test. In either case, a repeat COVID-19 test is not required. Likewise, a persistently positive test (if obtained) does not continue to exclude the patient should the other criteria be satisfied.
19. History of severe allergic, anaphylactic, or other hypersensitivity reactions to any of the study medications or their classes
20. Inability to swallow, retain and/or absorb oral medications
21. Pregnant or lactating or intending to become pregnant during the study interval
22. Other uncontrolled serious medical or psychiatric illness that would impact study participation and/or follow up in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To estimate the progression-free survival (PFS) benefit of fruquintinib in combination with TAS-102 as compared to fruquintinib | 24 months
  Progression free survival (PFS) defined as time from randomization to first observation of progression using RECIST v1.1 or death from any cause.

SECONDARY OUTCOMES:
Estimate the confirmed objective response rate (ORR) of fruquintinib in combination with TAS-102 as compared to fruquintinib | 24 months
  Objective response rate (ORR) defined as partial response or complete response using RECIST v1.1
Estimate the disease control rate (DCR) of fruquintinib in combination with TAS-102 as compared to fruquintinib | 24 months
  Disease control rate (DCR) defined as partial response, complete response, or stable disease using RECIST v1.1
Estimate the clinical benefit rate (CBR) of fruquintinib in combination with TAS-102 as compared to fruquintinib | 24 months
  Clinical benefit rate (CBR defined as the percentage of patients achieving a partial response, complete response, or stable disease for at least 6 months using RECIST v1.1
Estimate the overall survival (OS) of fruquintinib in combination with TAS-102 as compared to fruquintinib | 24 months
  Overall survival (OS) defined as time from randomization to death from any cause
Characterize the toxicity profile of fruquintinib in combination with TAS-102 | 24 months
  Toxicity profile comprised of: Incidence of grade 3 or more treatment-related adverse events (TRAE), Percent of patients requiring dose reductions or dose delays due to TRAE, Percent of patients requiring treatment discontinuation due to TRAE

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mount Sinai Cancer Research Program, Miami Beach, Florida
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: No